CLINICAL TRIAL: NCT05057559
Title: Prospective, Observational, Open-label, Clinical Investigation of Intra-articular Arthrosamid® Injection in Subjects With Knee Osteoarthritis
Brief Title: Observational Clinical Investigation of Arthrosamid in Knee Osteoarthritis
Acronym: LUNA
Status: Active, not recruiting | Type: Observational
Sponsor: Contura (Industry)
Responsible Party: Sponsor
Other Study IDs: CON-OA-002
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, long-term, observational, all-comers, open-label, multi-centre clinical investigation enrolling subjects with knee osteoarthritis who is eligible for treatment with Arthrosamid® according to the Instruction for Use.

DETAILED DESCRIPTION:
This is a prospective, long-term, observational, all-comers, open-label, multi-centre clinical investigation enrolling subjects with knee OA who is eligible for treatment with Arthrosamid® according to the Instruction for Use (IFU).

All subjects will be followed over an observational period of five years with yearly follow-up check points. The first follow-up visit should be six months after the treatment. All follow up visits can be performed as telephone visits.

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged ≥ 18 years
* Clinical diagnosis of knee OA

Exclusion Criteria:

* If an active skin disease or infection is present at or near the injection site
* If the joint is infected or severely inflamed
* If a degradable intra-articular injectable such as hyaluronic acid is present, it must be expected to be absorbed according to manufacturer's information for the specific product, before injection with Arthrosamid®
* If the patient has previously received treatment with a different non-absorbable injectable/implant
* If the patient has received a knee alloplasty or has any foreign material in the knee
* If the patient has undergone knee arthroscopy within the last 6 months
* If the patient has haemophilia or is in uncontrolled anticoagulant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from participating rheumatology or orthopedic centers.
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | 5 years
  The total number of treatment emergent adverse events

SECONDARY OUTCOMES:
WOMAC pain subscale | 6, 12, 24, 36, 48 and 60 months
  change from baseline in WOMAC (WOMAC Osteoarthritis Index) pain subscale
WOMAC stiffness subscale | 6, 12, 24, 36, 48 and 60 months
  change from baseline in WOMAC (WOMAC Osteoarthritis Index) stiffness subscale
WOMAC physical function subscale | 6, 12, 24, 36, 48 and 60 months
  change from baseline in WOMAC (WOMAC Osteoarthritis Index) physical function subscale
Patient's global assessment of impact of osteoarthritis | 6, 12, 24, 36, 48 and 60 months
  An eleven point, numeric rating scale (0-10) where 0 =" No impact" and 10 = "Worst imaginable impact"

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Tvinnemose, DVM., Study Chair — Contura
Locations (9):
- Denmark (2):
  - The Parker Institute, Copenhagen
  - Reumatolog i Odense, Odense
- France (2):
  - AP-HM hopitaux, Marseille
  - Clinique Saint Louis, Poissy
- Germany (2):
  - AmBeNet Hausarztpraxis, Leipzig
  - University Medical Center of Johannes Gutenberg-University Mainz (UMC-Mainz), Mainz
- Ospedale San Pietro Fatebenefratelli, Rome, Italy
- United Kingdom (2):
  - London North West University Healthcare, London
  - Royal Cornwall Hospital, Truro